CLINICAL TRIAL: NCT05490602
Title: Comparison Study in Different Sutures Techniques in Reduction of Known Abdominoplasty Complications and Improving Patients' Post-operative Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Socorro ORTIZ, Head of plastic surgery department, Brugmann University Hospital
Other Study IDs: CHUB-Raei Ahmad
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Abdominoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Running subcutaneous sutures technique: Abdominoplasty patients will be recruited. 50 patients will undergo the running subcutaneous sutures technique closures.
  Interventions: Procedure: Running subcutaneous sutures technique
- Classical closures: Abdominoplasty patients will be recruited. 50 patients will undergo classical closures.
  Interventions: Procedure: Classical closures

INTERVENTIONS:
Procedure: Running subcutaneous sutures technique — The Running subcutaneous sutures consist of running sutures in the profound and superficial dermis without knotting the thread (suture).
  Groups: Running subcutaneous sutures technique
Procedure: Classical closures — Classical closures
  Groups: Classical closures

SUMMARY:
After an important weight loss abdominoplasty has become one of the most frequent interventions to remove excess skin to achieve the best cosmetic and body perception psychological results after weight loss. The American Society of Plastic surgeons have published documents in 2004 indicating a 344% increase in the number of abdominoplasty cases.

Dog ears is one of the classical complications in body contouring and abdominoplasty which needs a scar revision to achieve the optimum cosmetic result. It's due to bad tension from the closed scar.

In a classical abdominoplasty wound closure subcuticular, (or intradermal) sutures can be interrupted or placed in a running fashion. Such a technique obviates the need for external skin sutures and circumvents the possibility of suture marks in the skin. Other techniques have been described in the literature to reduce abdominoplasty complication (seroma, hematoma, infection, dog ear, flap necrosis etc.. ) such as classical high lateral tension and lipo-aspiration on preventing dog ears and elongation scar was evaluated and progressive tension sutures. The running subcutaneous sutures that consist of running sutures in the profound and superficial dermis without knotting the thread(suture) showed less dog ears occurrence and other complications which leads to more patient satisfaction and less scar revision. Dog ear is referred to as a puckering of the skin that appears sometimes at the end of a scar, especially after procedures that involve some degree of skin tightening or when skin after the end of the scar is looser than skin along the scar itself creating a small excess of skin where the incision ends.

So far there's no reported epidemiology for dog ears in the literature, however it's mentioned in some papers where it's a common complication and reason for scar revision in abdominoplasty and breast reduction surgery.

The aim of this study is to compare the incidence of dog ear and other complications in classical abdominoplasty closure to running subcutaneous sutures, method, which decreases dog ear incidence, wound dehiscence, infection and hypertrophic scar which are actually quite common after abdominoplasty. This allows to avoid a scar correction surgery and have a better aesthetic outcome. The investigators also evaluate the amelioration of sexual activity after a pubis-pexy using SAQ(Sexual Activity Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

Adult women at our department undergoing primary abdominoplasty with transposition of umbilicus with or without liposuction

Exclusion Criteria:

* Age <18 or >65 years
* History of chemotherapy
* Smoker patient, diabetic patient
* Male patient
* < 6 months postpartum
* Non-compliant patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women at our department undergoing primary abdominoplasty with transposition of umbilicus with or without liposuction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of the wound | 1 year post surgery
  Pre-operative and post-operative photography will be taken in both groups allowing a visual assessment of the result. The end results will be examined by a third blinded party without a previous knowledge of which technique was used.
Pinch fat of dog ears | 3 months post surgery
  Absence/presence of dog ears. Dog ears is one of the classical complications in body contouring and abdominoplasty which needs a scar revision to achieve the optimum cosmetic result. It's due to bad tension from the closed scar.
Pinch fat of dog ears | 1 year post surgery
  Absence/presence of dog ears. Dog ears is one of the classical complications in body contouring and abdominoplasty which needs a scar revision to achieve the optimum cosmetic result. It's due to bad tension from the closed scar.
Sexual Activity questionnaire | 3 months post surgery
  The sexual activity questionnaire is a 20-item tool that is focused on the relational, emotional, and behavioral aspects of sexual activity in the general population. Each question is rated using a four-point Likert scale from 0 to 3 (0 : not at all, and 3 : very much)
Sexual Activity questionnaire | 1 year post surgery
  The sexual activity questionnaire is a 20-item tool that is focused on the relational, emotional, and behavioral aspects of sexual activity in the general population. Each question is rated using a four-point Likert scale from 0 to 3 (0 : not at all, and 3 : very much)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium